CLINICAL TRIAL: NCT03451552
Title: Patient Navigation in Primary Care and Access to Resources in the Community - A Randomized Controlled Trial
Brief Title: Patient Navigation in Primary Care and Access to Resources in the Community
Acronym: ARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other); University of Ontario Institute of Technology (Other); Laurentian University (Other); Bruyère Health Research Institute. (Other); Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20171215
Record Dates: First submitted 2018-01-11; First posted 2018-03-01 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Health Care Inequity, Patient Navigation
Keywords: Community Resources, Patient Navigator
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: This is a prospective, mixed method (patient) randomized controlled trial of navigation services provided by Ontario 211 vs. navigation services provided by a lay Patient Navigator. Randomization is 1:1 control:intervention.
  The mixed method design is a sequential, explanatory design. Patients having consented to participate in the study will complete a survey, after which their random assignment to one of two arms (intervention or control) will be revealed.
  The randomization schedule will be blocked at the practice level to ensure a balance of control and intervention patients for each practice, including all providers.
  Patients randomized to the intervention arm will have access to services provided by the ARC Patient Navigator, whereas patients randomized to the control arm will be directed to the Ontario 211 navigation service.
Masking Description: There is no masking in the study.The participant, their primary care provider, and the study team will know which arm the patient is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (211 services) (No Intervention): Patients allocated to the control arm will be directed to the Ontario 211 navigation service, which is already available to the general public free of charge. After consenting to participate in the study and completing the telephone survey, the research assistant will inform these patients that they can use existing navigation services provided by Ontario 211 to help them access the CR referred to them by their PHCP. The research assistant will instruct patients to dial 2-1-1 to obtain additional information on the nature of this service.
- Intervention (Patient Navigator) (Experimental): Patients allocated to the intervention arm will be offered the services of the ARC Patient Navigator. After consenting to participate in the study and completing the telephone survey, the research assistant will inform these patients that they can use the services offered by the ARC patient navigator to help them access the CR referred to them by their PHCP. Following a brief description of the services provided by the navigator (e.g., arrange transportation, make appointments, fill out forms, etc.), patients will be offered to be contacted by the navigator by telephone or to meet with the navigator in person on a day and time that is most convenient for them.
  Interventions: Behavioral: Patient Navigator

INTERVENTIONS:
Behavioral: Patient Navigator — Navigators will support patients to access community based resources for healthy living and self-management, rather than providing specific information about health issues. Navigators will teach patients how to identify available and relevant programs to meet their health-related goals, in their language of choice. The navigator will ensure that the individual understands the reason for referral and potential benefits. They will discuss social barriers potentially affecting patients' access to community health resources, and assist patients to prioritize their health goals and relevant resources to achieve these. The navigator will then assist patients to access the community-based services in the language of their choice to which they have been referred. The navigator may assist the patient in making appointments, coordinating transportation, and/or accompaniment to resources as required).
  Arms: Intervention (Patient Navigator)

SUMMARY:
Some people living with health problems require extra support to properly manage their conditions, as family doctors are only able to spend limited time in the office with these patients. There are many resources and programs in the community that can provide the necessary time and support for these patients, yet many patients are unaware that such resources exist. Patient navigators have been shown to be useful in helping patients with certain conditions (such as cancer) to get to the resources they need, especially when they have social challenges that make it difficult for them to reach these programs (for example, language or transportation barriers, poverty, or poor social support). This study will look at how helpful Navigators are to link patients at family doctors' offices to community resources. To do this, family doctors' offices in Ottawa and Sudbury will be recruited. All offices will receive training on directing patients to CRs and will be assigned a patient navigator to support patients access CRs. Half of the patients referred to CRs by their providers will have access to the navigator (intervention) assigned to the practice. This study will assess whether access to a navigator increases patients' access to community health and social services compared to usual standard of care. In addition, the study aims to understand whether English and French speaking individuals are as likely to benefit from a navigator in accessing community resources in the language of their choice.

DETAILED DESCRIPTION:
The proposed project builds on work conducted between 2013 and today. The Canadian Institutes of Health Research's Community Based Primary Health Care Team Grant SPOR initiative funded a five-year program of research (known as IMPACT: Innovative Models Promoting Access-to-Care Transformation, http://www.impactresearchprogram.com/). The goal of the IMPACT Project is to increase access to community-based primary health care for vulnerable populations. The lead for the Ontario arm of the IMPACT project, Simone Dahrouge, has undertaken a community engagement initiative within the Champlain Local Health Integration Network (LHIN) to understand the barriers patients face to adequately access community based health and social resources (CRs) and how these can be overcome. Under that funding, the team undertook an extensive consultation process to identify a regional priority gap, select and adapt an intervention, and implement and evaluate a single arm intervention. The investigators are currently in the last phase of that project, which is serving as a feasibility phase for the randomized controlled trial. The feasibility study is evaluating the acceptability, demand, implementation, adaption, integration, and practicality of the study intervention and related activities to optimize appropriate access to CRs for primary care patients. Enrolment for that project will be completed by March 2018. This study received ethics approval from the OHSN Research Ethics Board (Protocol #20160914-01H), Bruyère Continuing Care Research Ethics Board (Protocol #M16-1616-055), Hôpital Montfort Research Ethics Board (Protocol # SD-DP-27-02-17), and the University of Ottawa Research Ethics Board (Protocol # A05-17-04).That trial is a registered clinical trial: NCT03105635.

During the feasibility phase the team established a regional stakeholder advisory group (Champlain LHIN). The composition of the advisory group has been adapted to meet the needs of the study. In the initial phase the composition was broad until the region identified the priority area and approach to addressing the gap. The committee is now composed of patients of various minority communities who contribute their lived experience, primary care providers from different care models and leaders from organizations responsible for community services (Community Care Access Centres and Community Health Centres) who inform the feasibility of the approach for each context, and best approach to integrating of the two sectors, health planners (the LHIN Primary Care Lead, senior integration specialist and others) who bring their broader context health services knowledge as well as resources (such as practice transformation facilitation services) to the project, as well as other stakeholders that inform specific components of the intervention (Ontario 211, Champlain Healthline). That Committee meets regularly and contributes directly to the direction of the study design, implementation, evaluation and dissemination. Because the committee fundamentally represents the interests of the region, it is often referred to in this document as 'the region".

The initial consultative phase identified poor access to CRs as a priority access gap. The research team relied on a scoping review conducted for the IMPACT program and conducted several interviews and focus groups with community stakeholders to inform the best approach addressing this gap. The region selected to implement a patient navigator who can assist patients for whom the use of a community service is recommended by their primary care provider achieve access to that service. Primary care providers rarely make specific recommendations to access CRs; largely because they are unaware of these. They make general recommendations to improve healthy behaviours, but do not refer to specific types of services. Two realist reviews have been commissioned and completed by a team of experts to help us understand the critical success factors and shape our intervention. One review is focused on "community navigators" and the other on "primary care referral to community services" to help the team understand the factors that support us. This information was used to develop the ARC intervention. A number of themes identified in these reviews including training for clinical staff to identify and refer to relevant CRs to address patients' social barriers; implementing a champion within practice to integrate referral into usual care; use of electronic health records to prompt provider referral and share information between provider and the community; and developing a screening process and promotional material to prompt referral.

As a result, the region developed the Access to Resources in the Community/Accès aux Resources Communautaires (ARC) intervention. The ARC project will build on this work by focussing on improving access to community resources in patients' language of choice and emphasizing access to French-language resources for Francophones in Ontario.

PURPOSE

The purpose of this project is to optimize appropriate access to community based services for socially complex primary care patients, including Franco-Ontarians living in minority situations, and promote the continuity of information across primary and community care.

OBJECTIVES AND DELIVERABLES

Objective A: Optimize equitable utilization of community based resources

Deliverable 1: Effectiveness of a patient navigator on utilization of CRs

Deliverable 2: Make policy recommendations to address remaining gaps

Deliverable 3: Establish a model of navigation that is transferable and scalable.

Objective B: Support continuity of information across Primary and Community Care

Deliverable 4: Establish a process that support appropriate exchange of information across the two sectors

ELIGIBILITY:
There are 3 levels of participation in this study: primary care practices, primary care providers, and primary care patients.

1) Primary care practices

Inclusion criteria:

* Any practice providing comprehensive primary care services (i.e. excludes practices that provide walk in services only), except for Community Health Centres. This includes Reformed Fee For Service (Family Health Groups, Comprehensive Care Model), Capitation based models (Family Health Networks, Family Health Organizations), and interprofessional models (Family Health Teams)
* Located in a neighbourhood of the Champlain (Ottawa area) or North East (Sudbury area) LHIN that has a francophone population of 20% of greater, as listed identified in the Ottawa Neighbourhood Study and in custom neighbourhoods created by the city of Greater Sudbury for city planning purposes, both linked to Statistics Canada's 2011 Population Census, respectively.
* Having at least one primary care provider agreeing to participate in the study

Exclusion criteria:

* A Community Health Centre or clinics providing walk-in services only
* Practices that are under the traditional fee for service remuneration
* Located in a neighbourhood with less than 20% Francophone residents

Primary care providers:

Inclusion criteria:

* Work in a practice that meets the eligibility criteria participating practice will be invited to participate in the study.
* Is a Primary Health Care Provider: A health professional that may refer patients to CRs such as physicians, nurses, and social workers.

Exclusion criteria:

* None

Primary care patients:

Inclusion criteria:

* Patient identifies a primary care provider participating in the study as their main primary care provider
* Has received a recommendation for a CR from their PHCP
* Is able to communicate in English or French, or is willing to be served via a cultural interpreter/translator, preferably a family member.
* Is able to provide consent for the study (18 years of age or older), or has parental/guardian proxy to provide consent (minor patients, patients with cognitive deficits)

Exclusion criteria:

* Unable to provide consent and does not have a family member/guardian who can provide proxy consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Access to Community Resources | Three months
  The primary outcome measure is access to CRs amongst the patients participating in the study. This outcome reflects the ability of the navigator to help patients overcome barriers to access and reach the community resource. We will assess this outcome in both arms (control and intervention) three months after enrolment in the study through a patient survey. The outcome will be a count of the CRs accessed (as a patient may access more than one CR).

SECONDARY OUTCOMES:
Ability of the intervention to address equity | Baseline (i.e. the time of referrals (Pre-intervention) as well three months later, at the end of the patient three months intervention period
  Patient sociodemographic characteristics captured in the baseline survey (e.g. income, language, sex, age, immigration status) will be used to evaluate the intervention's success in supporting patients access the desired resource (main outcome variable) across various social strata.
Needs/Difficulties | Baseline (i.e. the time of referrals (Pre-intervention) as well three months later, at the end of the patient three months intervention period
  Section B in patient survey - related to ability to pay
Use of Healthcare | Baseline (i.e. the time of referrals (Pre-intervention) as well three months later, at the end of the patient three months intervention period
  Section B in patient survey - related to relationship with providers
Ability to engage | Baseline (i.e. the time of referrals (Pre-intervention) as well three months later, at the end of the patient three months intervention period
  Section C in the patient survey, one scale (including three concepts)
Quality of Life VR-12 | Baseline (i.e. the time of referrals (Pre-intervention) as well three months later, at the end of the patient three months intervention period
  Section F in patient survey
Health Action Process Approach | Time Frame: baseline (i.e. the time of referrals (Pre-intervention) as well three months later, at the end of the patient three months intervention period
  Section L in the patient survey - related to self efficacy and behaviour change
Patient Activation Measure | Baseline(i.e. the time of referrals (Pre-intervention) as well three months later, at the end of the patient three months intervention period
  Section M of patient survey - related to knowledge, confidence, and motivation to access services
Community service evaluation | Assessed after the three month patient intervention period.
  Section O in Patient Survey: used to evaluate whether the community service(s) were appropriate for the needs of the patient
Navigator Assessment (intervention arm only) | Assessed after the three month patient intervention period.
  An assessment of the Patient Navigator service received by patients in the intervention arm
Attitudes with reference to vulnerable populations | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  An assessment of primary care providers attitudes with reference to socially vulnerable populations
Practices with reference to vulnerable populations | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  An assessment of primary care providers practices with reference to socially vulnerable populations
Knowledge with reference to vulnerable populations | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  An assessment of primary care providers' Knowledge with reference to socially vulnerable populations
Contextual factors (e.g., organizational structure) | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  An assessment of the organization's (primary care organizations) organizational structure (section B of Provider survey)
Change valence | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  Section C of the provider survey
Change Climate | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  Section D of the provider survey
Organizational readiness for change | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  Section E of Provider Survey; An assessment of the organization's readiness to implement the navigator intervention
Implementation effectiveness | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  Section F of Provider SurveyAn assessment of the effectiveness of the navigator intervention within the primary care practice
Experience with the Navigator | Baseline(i.e. the time of referrals (Pre-intervention) and 10 months into the study intervention period.
  Section G of Provider Survey; An assessment of the providers' experience with the patient navigator, and how the intervention has affected their practice

CONTACTS AND LOCATIONS:
Overall Officials: Simone Dahrouge, PhD, Principal Investigator — Bruyère Health Research Institute.
Locations (1):
- Bruyere Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saluja K, Mahbub A, Gauthier AP, Lemonde M, Timony P, Durand F, Dahrouge S. Understanding patient barriers and enablers to accessing community resources: a qualitative study to inform navigation service delivery. BMC Prim Care. 2025 Oct 24;26(1):322. doi: 10.1186/s12875-025-03029-z. PMID 41136927

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03451552/Prot_SAP_000.pdf
  • Informed Consent Form: Practice and Provider Informed Consent Form (general) (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03451552/ICF_001.pdf
  • Informed Consent Form: Practice and Provider Informed Consent Form (interview) (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03451552/ICF_002.pdf
  • Informed Consent Form: Patient Informed Consent Form (general) (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03451552/ICF_003.pdf
  • Informed Consent Form: Patient Informed Consent Form (interview) (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03451552/ICF_004.pdf